CLINICAL TRIAL: NCT02493309
Title: The Impact of Cardio-respiratory Fitness on an Individual's Metabolic Response to Sitting and Light Activity Breaks
Brief Title: FIT 2 SIT - Are Metabolic Responses to Sitting/Light Breaks Mediated by Fitness?
Acronym: FIT2SIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 0458; CRN151741 (Other: Registry ID: UK Clinical Research Network)
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2014-10

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolonged sitting (Experimental)
  Interventions: Other: Prolonged sitting
- Light activity breaks (Active Comparator)
  Interventions: Other: Light activity breaks

INTERVENTIONS:
Other: Prolonged sitting — Condition A is referred to as the 'sitting' condition. Here participants will remain seated throughout the whole of the 7 ½ hour test period (8am - 3:30pm). On arrival, participants will have a cannula (a small tube that allows us to take blood) inserted into their arm; this will stay in the arm and allow us to take regular blood samples throughout the day. Blood samples and blood pressure will be taken at 30, 60, 120 and 180 minutes after breakfast. We will then provide a lunch meal and will continue taking blood samples and blood pressure at 30, 60, 120, 180 and 210 minutes after this lunch meal. In total, we will take 11 blood samples over the 7 ½ hour testing period.
  Arms: Prolonged sitting
Other: Light activity breaks — Condition B is the 'light activity breaks' condition. Participants will go through exactly the same process as condition A but will also be asked to do 5 minute bouts of slow walking on a treadmill every 30 minutes following breakfast and lunch. In total they will do 12 five minute walks on the treadmill throughout the 7 ½ hour test period (60 minutes of walking in total). In total, we will take 11 blood samples on the day.
  Arms: Light activity breaks

SUMMARY:
The purpose of this study is to determine whether an individuals cardio-respiratory fitness level can protect them from the negative metabolic impacts of prolonged sitting time.

Overall, it is hypothesised that in individuals with high fitness, the unfavourable effect of prolonged sitting (build up of sugar, fat and insulin in the blood following a meal) will not be as substantial, nor will light activity breaks be as advantageous, compared to individuals with lower fitness as they have a smaller scope for metabolic improvement.

DETAILED DESCRIPTION:
The FIT 2 SIT study requires three separate study visits in total.

At visit one, we will check the participants blood pressure, height, weight, waist measurement and body fat percentage, we will also take a blood sample to measure HbA1c and cholesterol, all of which will help confirm that this participant is eligible to continue in this study (some may be excluded based on results of the above). We will also measure the amount of energy participants expend per minute while at rest and during a slow walking task (3km.h on a treadmill) using a gas mask technique. Energy responses to sitting and walking differ between individuals, therefore it is of interest to observe how each participant in this study responds to these conditions as it may help explain any potential findings of this study. For instance, introducing walking breaks (by way of reducing sitting time) may only benefit those who have consequent increases in energy expenditure as a result of these breaks. Lastly, to mark the end of the first study visit, participants will be asked to perform an exercise test based on a treadmill to assess their fitness level. whilst running a special mask covering the nose and mouth will be worn to analyse breathing, this will be connected to a machine (gas analyser) that gives information on the amount of oxygen participants breathe in and out. The point at which the amount of oxygen they breathe in remains stable despite increases in exercise difficulty is the point that we will stop the exercise test because this tells us that they have reached their exercise capacity (called V02max), and from this we can determine fitness level.

Following this first visit we will have fitness level data from all participants. Recruiting participants with a diverse fitness level will then help to elucidate the role that an individuals fitness has on their response to the following treatment conditions.

Treatment condition A is referred to as the 'sitting' condition. Here participants will remain seated throughout the whole of the 7 ½ hour test period (8am - 3:30pm) whilst watching TV/DVD's, reading, using the internet, doing paperwork etc. at their will. On arrival, participants will have a cannula (a small tube that allows us to take blood) inserted into their arm; this will stay in the arm and allow us to take regular blood samples throughout the day, without the need for multiple needles. After we take the first blood sample, participants will sit quietly for an hour. We will then provide breakfast. Whilst sitting, we will take blood samples (using the cannula) and blood pressure at 30, 60, 120 and 180 minutes after breakfast. We will then provide a lunch meal and will continue taking blood samples and blood pressure at 30, 60, 120, 180 and 210 minutes after this lunch meal. In total, we will take 11 blood samples over the 7 ½ hour testing period. Although this may sound a lot, it is equivalent to around 8-9 teaspoons of blood over the course of the day.

Condition B is the 'light activity breaks' condition. Participants will go through exactly the same process as condition A but will also be asked to do 5 minute bouts of slow walking on a treadmill every 30 minutes following breakfast and lunch. In total they will do 12 five minute walks on the treadmill throughout the 7 ½ hour test period (60 minutes of walking in total). In total, we will take 11 blood samples on the day.

With data on each participants metabolic response to a meal during A) prolonged sitting and B) during an interrupted sitting condition, we can see how fitness influenced the results.

However, at present, the absence of laboratory randomised crossover trials assessing the 'extent' to which fitness moderates the relationship between sedentary behaviour and metabolic health markers appear absent from the literature, warranting further investigation, which is why this design was chosen.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Body Mass Index: 20 - 30 kg/m2
* Male and Female
* Aged: ≥ 25 to ≤ 55 years of age.
* Occupation: Work full-time in a predominantly sedentary occupation.

Exclusion Criteria:

Due to the nature of the trial, our exclusion criteria are as follows:

The participant may not enter the study if ANY of the following apply:

* Aged <25 or >55 years of age.
* Physical condition which limits full participation in the study
* Active psychotic illness or other significant illness which, in the view of the investigators, would prevent full participation
* Inability to communicate in spoken English
* Steroid use
* Known Type 2 Diabetes
* Pre-existing Cardio-vascular Disease (disease of the heart or blood vessels at present or in the past) For example: Heart attack, Stroke or Angina.
* Pregnancy
* Smoker
* Terminal illness

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Blood glucose Area Under the Curve (AUC) | Assessed via 11 blood samples throughout each treatment condition throughout the 7.5 hour period
  Blood glucose AUC refers to the spike of an individuals blood sugar following a meal, the aim of which is to reduce the spike and consequently reduce the area under the curve.

SECONDARY OUTCOMES:
Blood Triglyceride AUC | Assessed via 11 blood samples throughout each treatment condition throughout the 7.5 hour period
  Refers to an individuals triglyceride response to a meal over a prolonged time period during each treatment.
Insulin AUC | Assessed via 11 blood samples throughout each treatment condition throughout the 7.5 hour period
  Refers to an individuals insulin response to a meal over a prolonged time period during each treatment.
Blood Pressure | Taken immediately before each blood sample is taken.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Yates, PhD, Principal Investigator — University of Leicester
Locations (1):
- Leicester Diabetes Centre, Leicester General Hospital, Leicester, Leicestershire, United Kingdom

REFERENCES:
- See also: NIHR Leicester-Loughborough Diet, Lifestyle and Physical Activity Biomedical Research Unit — http://www.ll.dlpa.bru.nihr.ac.uk/
- See also: Leicester Diabetes Centre — http://www.leicesterdiabetescentre.org.uk/